CLINICAL TRIAL: NCT06065878
Title: Comparison Of The Analgesic Efficacy Of IPACK (Interspace Between The Popliteal Artery And Capsule Of The Posterior Knee) Block Alone And IPACK Block Combined With Genicular Block In Patients Planned For Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cenk Gacemer (Other)
Responsible Party: Sponsor-Investigator, Cenk Gacemer, Principal Investigator, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPACKvsIPACK&GNB
Record Dates: First submitted 2023-09-04; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pain, Joint; Knee Arthropathy; Anesthesia; Orthopedic Disorder
Keywords: IPACK Block; Genicular Nerve Block; Total Knee Arthroplasty
MeSH Terms: conditions — Arthralgia; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPACK block (No Intervention): In the IPACK block group, a 20 mL solution containing 50 mg of 0.25% bupivacaine (Buvicaine®, Polifarma, Tekirdağ, Turkey) and 8 mg of dexamethasone (Dekort®, Deva, Istanbul, Turkey) was infiltrated between the popliteal artery and femur, starting 2 cm distal to the popliteal artery and being withdrawn while infiltrating proximally.
- IPACK + Genicular Nerve Block (Active Comparator): In the IPACK+GNB group, 12 mL of the same solution was used for the IPACK block infiltration. Then, the patient was positioned supine, and an ultrasound (Logiq e®, GE, Boston, USA) linear probe was placed approximately 2-3 cm above the patella, in the midline of the femur, with a sagittal plane angle of 45 degrees to visualize the femur and genicular artery . The visible needle was advanced in-plane towards the genicular artery, and 4 mL of local anesthetic solution was injected on the surface of the femur. The same procedure was repeated for the superior lateral genicular nerve block, creating a mirror image on the lateral side of the femur.
  Interventions: Procedure: IPACK + Genicular Nerve Block

INTERVENTIONS:
Procedure: IPACK + Genicular Nerve Block — IPACK and Genicular Nerve block were applied with the same total volume of local anesthetic as the control group.
  Arms: IPACK + Genicular Nerve Block

SUMMARY:
The IPACK (interspace between the popliteal artery and capsule of the posterior knee) block is a regional anesthesia technique in which a local anesthetic is infiltrated under ultrasound guidance between the popliteal artery and the capsule of the posterior knee. This technique blocks the branches of the obturator nerve, the common peroneal nerve, and the tibial nerve in the popliteal region. In the context of knee arthroplasty, the application of the IPACK block has been associated with lower scores for ambulatory pain, lower scores for resting pain, and reduced morphine consumption .

The genicular nerves, including the superomedial, inferomedial, superolateral, inferolateral genicular nerves, and the infrapatellar branch of the saphenous nerve, comprise the five main innervation branches of the knee. Clinically, they play an important role in the anterior sensory innervation of the knee.

In the study, the investigators aimed to prospectively, double-blind, and randomly compare the postoperative analgesic efficacy of combined IPACK block and genicular block with the sole application of IPACK block in patients undergoing total knee arthroplasty (TKA). The investigators hypothesized that in blocks performed with equal volumes, there might be a spread of the local anesthetic solution from the IPACK block area to the genicular block area, and the investigators investigated this hypothesis.

DETAILED DESCRIPTION:
Chronic knee pain, observed in the range of 7-33% in the society, is often caused by osteoarthritis. The knee joint consists of four bones: the femur, tibia, the largest sesamoid bone called the patella, and the fibula, although it does not directly join the joint. It is divided into three compartments called the medial tibiofemoral, lateral tibiofemoral, and patellofemoral, which share a common synovial cavity. Additionally, the knee joint is composed of the patellofemoral and tibiofemoral joints. The knee joint is supported by ligaments that provide stability and muscles and tendons that maintain its dynamic structure.

The superomedial quarter of the anteromedial aspect of the knee joint is innervated by the nervus vastus medialis, the medial branch of the nervus vastus intermedius, and the superior medial genicular nerve. The inferomedial quarter is innervated by the infrapatellar branch of the saphenous nerve and the inferior medial genicular nerve. The superolateral quarter of the anterolateral aspect is innervated by the nervus vastus lateralis, the lateral branch of the nervus vastus intermedius, the superior lateral genicular nerve, and the articular branches of the common fibular nerve. The inferolateral portion is innervated by the inferior lateral genicular nerve and the recurrent fibular nerve. The posterior sensation of the knee is provided by the popliteal plexus. Due to the dense innervation of the knee joint, approximately 60% of patients undergoing knee prostheses experience severe pain, while 30% describe a moderate level of pain.

The IPACK (interspace between the popliteal artery and capsule of the posterior knee) block is a regional anesthesia technique in which a local anesthetic is infiltrated under ultrasound guidance between the popliteal artery and the capsule of the posterior knee. This technique blocks the branches of the obturator nerve, the common peroneal nerve, and the tibial nerve in the popliteal region. In the context of knee arthroplasty, the application of the IPACK block has been associated with lower scores for ambulatory pain, lower scores for resting pain, and reduced morphine consumption .

The genicular nerves, including the superomedial, inferomedial, superolateral, inferolateral genicular nerves, and the infrapatellar branch of the saphenous nerve, comprise the five main innervation branches of the knee. Clinically, they play an important role in the anterior sensory innervation of the knee. GNB (genicular nerve block) and radiofrequency ablation techniques are utilized in the treatment of chronic osteoarthritis and have recently gained popularity in postoperative pain management following knee surgeries.

In our study, the investigators aimed to prospectively, double-blind, and randomly compare the postoperative analgesic efficacy of combined IPACK block and genicular block with the sole application of IPACK block in patients undergoing total knee arthroplasty (TKA). The investigators hypothesized that in blocks performed with equal volumes, there might be a spread of the local anesthetic solution from the IPACK block area to the genicular block area, and the investigators investigated this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral total knee arthroplasty
* Between the ages of 18 and 80,
* Classified as American Society of Anesthesiologists (ASA) class I-III

Exclusion Criteria:

* Patients under 18 years old or over 80
* ASA scores IV and above,
* pregnant or suspected of being pregnant,
* allergic to local anesthetics,
* coagulopathy,
* injection site infection,
* significant neurological or psychiatric disorders,
* severe cardiovascular diseases,
* chronic opioid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Scores- Visual Analog Scale scores | Postoperatively 0 minute, 30th minute , 60th minute , 2nd hour, 4th hour, 8th hour, 12th hour and 24th hour
  Visual Analog Scale scores. 0 to 10 scale. 0 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
Time to First Analgesic Requirement | Postoperative 24 hours
  the time to first rescue analgesic requirement was recorded and referred to as the analgesic time
Patient and Surgeon Satisfaction- 5 point Likert scale | Postoperative 24th hour.
  5 point Likert scale is from 1 to 5. 1 is Very Dissatisfied, 5 is very Satisfied.
Mobilization Time | Postoperative 24 hours
  The time elapsed until the patient could stand up and start walking with or without support was recorded as the mobilization time

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A. Fırat, K. Başarır, and M. Binnet, Türk Ortopedi ve Travmatoloji Birliği Derneği Diz ekleminin cerrahi anatomisi, TOTBİD Dergisi, 2011; 10 (1): 38-44
- [Background] GARDNER E. The innervation of the knee joint. Anat Rec. 1948 May;101(1):109-30. doi: 10.1002/ar.1091010111. No abstract available. PMID 18915634
- [Background] Seo SS, Kim OG, Seo JH, Kim DH, Kim YG, Park BY. Comparison of the Effect of Continuous Femoral Nerve Block and Adductor Canal Block after Primary Total Knee Arthroplasty. Clin Orthop Surg. 2017 Sep;9(3):303-309. doi: 10.4055/cios.2017.9.3.303. Epub 2017 Aug 4. PMID 28861197
- [Background] Xiumei T, Yahao L, Siwei D, Ning N. Correction: Analgesic efficacy of adding the IPACK block to multimodal analgesia protocol for primary total knee arthroplasty: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2022 Dec 26;17(1):565. doi: 10.1186/s13018-022-03460-3. No abstract available. PMID 36572894
- [Background] Kukreja P, Venter A, Mason L, Kofskey AM, Northern T, Naranje S, Ghanem E, Lawson PA, Kalagara H. Comparison of Genicular Nerve Block in Combination With Adductor Canal Block in Both Primary and Revision Total Knee Arthroplasty: A Retrospective Case Series. Cureus. 2021 Jul 29;13(7):e16712. doi: 10.7759/cureus.16712. eCollection 2021 Jul. PMID 34471571
- [Background] Roberts SL, Stout A, Dreyfuss P. Review of Knee Joint Innervation: Implications for Diagnostic Blocks and Radiofrequency Ablation. Pain Med. 2020 May 1;21(5):922-938. doi: 10.1093/pm/pnz189. PMID 31407791
- [Background] Elsaman AM, Maaty A, Hamed A. Genicular nerve block in rheumatoid arthritis: a randomized clinical trial. Clin Rheumatol. 2021 Nov;40(11):4501-4509. doi: 10.1007/s10067-021-05821-5. Epub 2021 Jul 2. PMID 34213672
- [Background] Tran J, Giron Arango L, Peng P, Sinha SK, Agur A, Chan V. Evaluation of the iPACK block injectate spread: a cadaveric study. Reg Anesth Pain Med. 2019 May 6:rapm-2018-100355. doi: 10.1136/rapm-2018-100355. Online ahead of print. PMID 31061110